CLINICAL TRIAL: NCT05455281
Title: A Pilot, Observational, Prospective Study to Evaluate the Performance of CHLOE Algorithm on the Prediction of Blastocyst Formation in Women Undergoing In-vitro Fertilization
Brief Title: Performance of CHLOE Algorithm on the Prediction of Blastocyst Formation
Acronym: CHLOE
Status: Completed | Type: Observational
Sponsor: Fairtility (Industry)
Responsible Party: Sponsor
Other Study IDs: FRT-01-22
Record Dates: First submitted 2022-06-29; First posted 2022-07-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: CHLOE — CHLOE is designed to automatically analyze events related to embryo development from Time Lapse Incubator (TLI) images and provide prediction on the likelihood of embryos developing to the blastocyst. This information can assist embryologists and IVF professionals in the selection of the most viable embryo for transfer or freezing, when there are multiple embryos deemed suitable.

SUMMARY:
This is an observational, prospective, single-arm, multi-center, clinical study to evaluate the performance of CHLOE, an Artificial Intelligence (AI)-based software application, as adjunct information to support identifying embryos on Day 3 that are most likely to form blastocysts.

DETAILED DESCRIPTION:
The study is an observational, prospective, single-arm, multi-center, clinical study in order to evaluate the performance of CHLOE, an Artificial Intelligence (AI)-based software application, as adjunct information to support identifying embryos on Day 3 that are most likely to form blastocysts on Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh IVF treatment using their own eggs
* At least 18 years of age
* Total antral follicle count (AFC) of at least 12 as measured by ultrasound prior to stimulation (in cases where AFC is performed)
* Basal day 3 follicle-stimulating hormone levels (FSH) < 10 IU
* At least 8 normally fertilized eggs at pronuclear (2PN) stage
* Fertilization using only ejaculated sperm (fresh or frozen) - no surgically removed sperm
* At least 2 cells embryo
* At least part of the embryos were cultured until Day 5 (i.e., 114-116 hours)
* IVF treatment cycles were performed during 2020-2021

Exclusion Criteria:

* Use of re-inseminated eggs
* Embryos that underwent day 3 biopsy for preimplantation genetic testing (PGT)
* Gestational carriers
* Concurrent participation in another clinical study
* Previous enrollment in this clinical study (i.e., previous cycles of the same women)
* History of cancer
* Embryos that underwent biopsy at cleavage stage

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing IVF
Study Population: Women undergoing fresh IVF treatment
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
The association between the adjunct prediction using CHLOE of blastocyst outcome and the actual blastocyst outcome for a subset of good/fair embryos | 3 days
  The prediction of blastocyst outcome using CHLOE algorithm, and the actual blastocyst outcome for a subset of good/fair embryos will be measured using odds ratio.

SECONDARY OUTCOMES:
The association between the adjunct prediction using CHLOE of blastocyst outcome and the actual blastocyst outcome for all embryos | 3 days
  The prediction of blastocyst outcome using CHLOE algorithm, and the actual blastocyst outcome for all embryos will be measured using odds ratio.
Blastocyst formation using traditional human morphology only for all embryos | 3 days
  The prediction of blastocyst outcome using traditional human morphology only, and the actual blastocyst outcome for all embryos will be measured using odds ratio.
Blastocyst formation based on the CHLOE algorithm prediction for a subset of good/fair embryos | 3 days
  The prediction of blastocyst outcome using the CHLOE algorithm for each individual embryologist will be measured using odds ratio for a subset of good/fair embryos.

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Gilgun-Sherki, PhD, MBA, Study Director — Head of Clinical and Regulatory Affairs
Locations (3):
- United States (2):
  - IVF Florida, Margate, Florida
  - Mayo clinic, Rochester, Minnesota
- Hadassah University Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No